CLINICAL TRIAL: NCT05885919
Title: Effect of Early Versus Late Initiation of Edaravone Dexborneol on Neural Function in Patients With Acute Ischemic Stroke-A Multicenter, Randomized, Double-blind, Placebo-controlled, Trial
Brief Title: Effect of Early Versus Late Initiation of Edaravone Dexborneol on Neural Function in Patients With Acute Ischemic Stroke
Acronym: EARLYS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Shenjingneike
Record Dates: First submitted 2023-05-14; First posted 2023-06-02 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-04

CONDITIONS: Ischemic Stroke, Acute; Treatment Outcome
Keywords: Acute ischemic stroke; Semi-dark band; Brain cell protection; Time window; Erafurone dextrol injection; Treatment Outcome
MeSH Terms: conditions — Ischemic Stroke | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Subjects with AIS who met the criteria for inclusion were stratified 1:1 from onset to use of the investigational drug: early (< 3 hours) and late (3-6 hours).
  Each layer was then randomly assigned to two groups in a 1:1 ratio: the right group and the placebo group.
  Test group:
  Edaravone dextronicol concentrated solution for injection, 15ml / time (37.5mg / time, of which edaravone 30mg, (+)-2-camphol 7.5mg), that is, 3 bottles / time, 2 times a day, for 12±2 days;
  Control group:
  Equal dose of placebo, 15 ml / time, that is, 3 sticks / time, 2 times a day for 12±2 days.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edaravone Dexborneol group (Experimental): Patients in this arm will be given Edaravone Dexborneol Concentrated Solution for injection twice a day for 10 to 14 days.
  Interventions: Drug: Edaravone Dexborneol Concentrated Solution for injection
- Edaravone Dexborneol Placebo group (Placebo Comparator): Patients in this arm will be given a placebo of Edaravone Dexborneol for injection twice a day for 10 to 14 days
  Interventions: Drug: Edaravone Dexborneol placebo

INTERVENTIONS:
Drug: Edaravone Dexborneol Concentrated Solution for injection — Edaravone and Dexborneol Concentrated Solution for Injection, 15 ml (37.5 mg, containing edaravone 30 mg and dexborneol 7.5 mg) in 3 ampoule bottles, twice a day for 10 to 14 days.
  Other Names: Xian Bi Xin,CFDA Approval Number H20200007
  Arms: Edaravone Dexborneol group
Drug: Edaravone Dexborneol placebo — Edaravone and Dexborneol placebo, 15 ml in 3 ampoule bottles, twice a day for 10 to 14 days.
  Other Names: Xian Bi Xin placebo
  Arms: Edaravone Dexborneol Placebo group

SUMMARY:
The primary objective of this study was to evaluate the efficacy and safety of initiation of edaravone dextivel therapy compared with placebo in patients with acute ischaemic stroke (early and late) and to explore the optimal time window for "brain cell protective therapy" of edaravone dexborneol.

DETAILED DESCRIPTION:
This is a multicentre, randomized, double-blind, placebo-controlled trial that aims to investigate the efficacy and safety of (early and late) initiation treatment of Edaravone Dexborneol versus placebo in patients with acute ischemic stroke, and to explore the optimal time window for "brain cell protective therapy" of Edaravone Dexborneol. Patients who were eligible to the inclusion criteria and ineligible to the exclusion criteria will be stratified by time to trial drug: early (<3 hours) and late (3-6 hours). Then each layer will be randomly assigned into two groups by a 1:1 ratio after the ICF was received. Patients in one arm will be given 15ml edaravone and dexborneol concentrated solution for injection (37.5mg, containing edaravone 30mg and dexborneol 7.5mg) twice a day for 10-14 days, and those in the other arm will be given an equivalent placebo drug. All patients will be followed up for 90 days. The primary outcome is the proportion of modified Rankin Scale 0-2 and the safety outcome is the proportion of severe adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old, gender is not limited;
* Clinically confirmed acute ischemic stroke;
* Within 6 hours of the onset of this stroke;
* NIHSS score of 4-24 at enrollment;
* mRS score before onset≤ 1 point;
* Subject and subject's agent are able and willing to sign informed consent.

Exclusion Criteria:

* CT indicates intracranial hemorrhagic diseases, such as hemorrhagic stroke, subdural hematoma, ventricular hemorrhage, or subarachnoid hemorrhage, etc.;
* Previously known severe liver or kidney insufficiency (ALT or AST is greater than 3.0×ULN; serum Creatinine (SCr) is greater than 1.5×ULN, Creatinine Clearance (CrCl) is less than 50 ml/min or dialysis;
* Systolic blood pressure≥220 mmHg or <90mmHg；
* Recent stroke within prior 1 month；
* Hypersensitive to edaravone, (+)-2- dexborneol or auxiliary materials;
* Prior receipt of edaravone or any other neuroprotective drugs;
* History of congenital or acquired hemorrhagic disease, coagulation factor deficiency disease, or thrombocytopenic disease, etc.;
* Pregnancy, lactation, or planned pregnancy within 90 days;
* Those who cannot complete informed consent or follow-up treatment due to severe mental disorder or dementia;
* Those with a malignant tumor, severe systemic diseases, or predict survival time <90 days;
* Participate in another interventional clinical study within 30 days before randomization or participate in another interventional clinical study;
* The investigators consider the patients are not suitable for this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
A 90-day mRS score of 0 to 2 in participants with acute ischaemic stroke | 90 days
  To assess the proportion of participants (early and late) who started edaravone dextrol compared with placebo with a 90-day mRS score of 0 to 2 in participants with acute ischaemic stroke

SECONDARY OUTCOMES:
Neurological recovery | 90 days
  The difference value of the NIHSS between Day 14/Day 90 and the baseline.
Modified Rankin scale | 90 days
  used to evaluate the functional outcomes after AIS，good prognosis (mRS score 0-2), generally good prognosis (mRS score 3-4) , Poor prognosis (mRS >4 points).
Quality of life score (EQ-5D) | 90 days
  Generic health status evaluated by EQ-5D questionnaire at the end of the therapy.
The incidence of serious adverse events | 90 days
  The percentage of the Severity Adverse Events within the 14 days/90 days of the therapy.
All-cause mortality | 90 days
  All-cause mortality at 90 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Le, PhD, Principal Investigator — Department of Neurology，XiangYa School of Medicine
Locations (3):
- China (3):
  - Brain Hospital of Hunan Province, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - XiangYa School of Medicine, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xu J, Wang A, Meng X, Yalkun G, Xu A, Gao Z, Chen H, Ji Y, Xu J, Geng D, Zhu R, Liu B, Dong A, Mu H, Lu Z, Li S, Zheng H, Chen X, Wang Y, Zhao X, Wang Y; TASTE Trial Investigatorsdagger. Edaravone Dexborneol Versus Edaravone Alone for the Treatment of Acute Ischemic Stroke: A Phase III, Randomized, Double-Blind, Comparative Trial. Stroke. 2021 Mar;52(3):772-780. doi: 10.1161/STROKEAHA.120.031197. Epub 2021 Feb 16. PMID 33588596
- [Result] GBD 2019 Stroke Collaborators. Global, regional, and national burden of stroke and its risk factors, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Neurol. 2021 Oct;20(10):795-820. doi: 10.1016/S1474-4422(21)00252-0. Epub 2021 Sep 3. PMID 34487721